CLINICAL TRIAL: NCT06258759
Title: The Effects of Autologous Platelet-rich Plasma Supplement During Sperm Cryopreservation
Brief Title: The Effects of Autologous Platelet-rich Plasma Supplement During Sperm Cryopreservation on Post-cryopreserved Sperm Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 151/2566
Record Dates: First submitted 2023-12-22; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Autologous Platelet-rich Plasma Supplement; Sperm Cryopreservation; Post-cryopreserved Sperm Quality; Semen Analysis
Keywords: Sperm; Platelet rich plasma; Vitrification; Cryopreservation; Semen analysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental: semen (Experimental): a semen of normal semen analysis
  Interventions: Biological: autologous platelet-rich plasma supplement
- placebo: semen (Experimental): a semen of normal semen analysis
  Interventions: Biological: no autologous platelet-rich plasma supplement

INTERVENTIONS:
Biological: autologous platelet-rich plasma supplement — the semen of the additional autologous platelet-rich plasma supplement group will be added by 5% PRP and mixed with Sperm Freezing Medium and undergo cryopreservation by Sperm vitrification for 14 days
  Arms: experimental: semen
Biological: no autologous platelet-rich plasma supplement — the semen mixed with Sperm Freezing Medium and undergo cryopreservation by Sperm vitrification for 14 days
  Arms: placebo: semen

SUMMARY:
Sperm cryopreservation is an essential procedure for male fertility in certain situations, like cancer, vasectomy or other obstructive surgeries, autoimmunity diseases, immunosuppressive therapeutic strategies, or when the male partner is incapable of providing sufficient spermatozoa on the day of egg retrieval. Semen cryopreservation is mainly associated with decreased viability, motility, and DNA damage of spermatozoa due to the osmotic and mechanical stresses attributed to the freezing-thaw- ing process. Sperm cryodamage mainly originates from osmotic changes, cold shock, intracellular ice crystal formation, and oxidative stress. Based on this, some protective strategies have been proposed and developed, even the addition of cryoprotectants. Recently, Platelet-rich plasma (PRP) is becoming very popular in medicine. The therapeutic effect of platelets is related to alpha granule contents. A study showed that PRP modulates ROS toxicity through a different mechanism. VEGF detoxify oxidative damage via activation of the nuclear factor (erythroid- derived 2)-like2 (Nrf2) pathway. Oxidative stress modulation and apoptosis inhibition both have an essential role during the cryopreservation process. In this case, it raises the question of whether PRP can improve the sperm quality against freeze-thawing-induced damage. Therefore, the present study aimed to examine different concentrations of PRP on frozen-thawed sperm parameters of vitality, morphology, motility and DNA fragmentation

DETAILED DESCRIPTION:
* Each participant will be collected a semen and PRP.
* Each semen will be separated into two specimens as the additional autologous platelet-rich plasma supplement group and control group (no adding autologous platelet-rich plasma). Both groups will undergo cryopreservation by Sperm vitrification for 14 days.
* The additional autologous platelet-rich plasma supplement group: the semen will be added by 5% PRP and mixed with Sperm Freezing Medium and undergo cryopreservation by Sperm vitrification for 14 days.
* The control group (no adding autologous platelet-rich plasma): the semen will be mixed with Sperm Freezing Medium and undergo cryopreservation by Sperm vitrification for 14 days.
* After 14 days, the vitrified semen was transferred to a water bath of 37 °C for thawing. And analyzed Semen analysis via Computer Assisted Sperm Analysis: CASA and analyzed DNA fragmentation

ELIGIBILITY:
Inclusion Criteria:

1. A man who be a Rajavithi hospital clients or staff.
2. Aged 20-40 years old.
3. Has normal semen analysis.
4. Can communicate and understand Thai language very well.
5. Voluntarily participated in the research.
6. Sexual abstinence for 2-7 days.

Exclusion Criteria:

1. A man who ever diagnosed with infertile patient.
2. A wan who diagnosed with any hematological disease such as Coagulation disorders, Hypertension, Thrombocytopenia, Platelet dysfunction.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sperm vitality | 14 days after cryopreservation
  Sperm vitality (percentage) after thawing

SECONDARY OUTCOMES:
Sperm motility | 14 days after cryopreservation
  Sperm motility (percentage) after thawing
Sperm morphology | 14 days after cryopreservation
  Sperm morphology (percentage of normal form) after thawing
DNA fragmentation | 14 days after cryopreservation
  DNA fragmentation (percentage) after thawing

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
drafting official document and distribute to IPD about study protocal, statistical analysis plan. inform consent and clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR